CLINICAL TRIAL: NCT00646243
Title: Italian Multicenter PROject on Echo Assessment of Left VEntricular (IMPROVE) Dyssynchrony Study
Brief Title: Echo Assessment of Intraventricular Dyssynchrony
Acronym: IMPROVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Italian Society of Cardiology (Other)
Responsible Party: Luigi P. Badano, M.D., Ospedale Universitario di Udine
Other Study IDs: IMPROVE
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Heart Failure; Ischemic Heart Disease; Dilated Cardiomyopathy
Keywords: Heart failure; echocardiography; cardiac resynchronization therapy; left ventricular dyssynchrony
MeSH Terms: conditions — Myocardial Ischemia; Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Heart Failure: 216 consecutive consenting patients with refractory heart failure candidate to cardiac resynchronization therapy by clinical and electrocardiographic criteria
- 2 Healthy subjects: 120 healthy subject includes defined as absence of history and symptoms of any cardiovascular disease, normal physical examination and ECG.

SUMMARY:
Background. Clinical benefits of cardiac resynchronization therapy (CRT) have been clearly demonstrated in heart failure (HF) patients with severe left ventricular (LV) dysfunction and wide QRS at surface electrocardiogram. However, there is a growing evidence that QRS duration poorly predicts responses to CRT, and that ~30% of patients do not experience any benefit from CRT when pre-implant dyssynchrony is defined according to electrocardiographic criteria. A number of echocardiographic criteria have been proposed to assess mechanical LV dyssynchrony, but at present there is no consensus on their use to predict response to CRT.

Study Design. The Italian Multicenter PROject on echo assessment of left VEntricular (IMPROVE) dyssynchrony study is a prospective, multicenter, observational study aimed to assess feasibility and predictive power of mechanical dyssynchrony assessed by echocardiography in consecutive consenting patients candidate to CRT by clinical and electrocardiographic criteria. IMPROVE will enroll 120 healthy subjects and 216 HF patients in 6 sites in Italy. CRT response criteria will be based on improvement in NYHA class and LV reverse remodeling evaluated by 3D-echocardiography. Enrollment is expected to conclude early 2009.

Implications. CRT is today part of the therapeutic armamentarium for symptomatic HF patients refractory to medical therapy, with wide QRS complex and severe LV systolic dysfunction. The IMPROVE study has been designed to evaluate reference values of indexes of ultrasound mechanical dyssynchrony that have been proposed in the literature and compare their ability to predict response to CRT in HF patients.

DETAILED DESCRIPTION:
The IMPROVE study has 3 main purposes:

1. definition of reference values of echocardiographic mechanical dyssynchrony (DYS) indexes in a population of healthy subjects;
2. definition of the feasibility and reproducibility of such indexes in healthy subjects and in HF patients undergoing implantation of a biventricular pacemaker;
3. definition of the accuracy of such indexes for predicting response to CRT.

   STUDY DESIGN. Multicenter, prospective, observational study that will be carried out in 6 Italian sites of acknowledged expertise in LV DYS evaluation and biventricular pacemaker implantation. At least 120 healthy subjects (about 20 per site) and 216 HF patients candidates to CRT (about 36 per site) will be enrolled. With this sample volume it is possible to test statistically significative differences of about 7%, with an alfa=0.05 and beta=0.50. Definition of healthy subject includes absence of history and symptoms of any cardiovascular disease, normal physical examination and ECG. The same commercial ultrasound equipment will be used for image acquisition in each investigating center and echo studies will be sent to a core-lab for analysis.

   Both ischemic and non ischemic etiology of HF will be considered. Patients with permanent or persistent atrial fibrillation or flutter will be excluded, as these patients cannot benefit from the atrial-ventricular component of resynchronization.

   The following evaluations:

   - clinical examination, including NYHA class estimate;
   * 12-lead standard ECG;
   * echocardiographic examination. will be performed within 7 days before CRT and repeated after 3 months of CRT. Patients will receive all appropriate treatments for HF, which include a diuretic, an ACE- inhibitor, or an angiotensin receptor blocker and usually digitalis and a beta-blocker. Doses of these background medications will be kept maximized during the follow-up period.

   Response to CRT will be assessed after 3 months of CRT as follows:
   * CRT response: combined end-point defined as NYHA class improvement by at least one grade and echocardiographic LV end-systolic volume decrease by at least 10% with respect to baseline (variations are considered as relative values);
   * CRT non-response: death for cardiac causes or failure to reach the above pre-specified NYHA class and echocardiographic changes.

   Patients who will die for non-cardiac causes will not be considered as non-responders but will exit the study.

   ECHOCARDIOGRAPHY

   - Image acquisition. Conventional M-mode and B-mode two-dimensional (2D) echocardiography, conventional pulsed (PW), continuous (CW) wave and color Doppler, tissue Doppler imaging (TDI), triplane tissue synchronization imaging (TSI) and RT3DE techniques will be used for data acquisition in each site using a GE-Vingmed Vivid 7 Dimension echo scanner (GE Healthcare, Horten, Norway), equipped with a broad-band M3s probe (2.5 MHz) and a matrix-array 3V probe (2.5 MHz), and the EchoPAC software v. BT05 or more.

   Ultrasound scanning will be performed after 10 min rest with the patient in left lateral decubitus position (unless differently specified). Standard parasternal, apical and subcostal views will be acquired in conventional 2D modality. From the parasternal approach the 3 standard short-axis views (basal, mid-ventricle and apical) will be collected. The mid-LV short-axis view will be selected with the papillary muscle as a consistent internal anatomic landmark, and great care will be taken to orient the image to the most circular geometry possible. Oblique views with elliptical geometry will not be recorded. From the apical approach, the 3 standard apical views (4-chamber, 2-chamber, long-axis) will be acquired also in triplane mode. Using this technique, once the apical 4-chamber view is optimized similar to the one obtained with the traditional 2D transducer, secondary image planes (i.e., apical 2-chamber and long-axis views) are automatically displayed in a quad screen view. The relative angles between the 3 image planes will be adjusted to acquire the 3 standard apical views according to anatomical landmarks. All apical images (2D and triplane) will be collected in gray-scale, color TDI and TSI modality. Gain settings will be adjusted for routine clinical gray-scale 2D imaging to optimize endocardial definition; frame rates will be kept between 55 and 70 fps to allow subsequent speckle tracking analysis (see below). Sector angle, depth, and Doppler pulse repetition frequency will be optimized to obtain the highest possible frame rate (>100 fps) avoiding loss of spatial data and aliasing in the TDI modality. RT3DE datasets will be obtained from the apical approach immediately after acquisition of 2D apical views, with the patient in the same position. In order to include the entire LV into the 3D dataset, a full-volume acquisition mode will be used. Using this approach it is possible to "stitch" together 4 sub-volumes obtained in real-time over consecutive cardiac cycles according to a previously described technique and protocol. This will create an on-line rendered image of the scanning sector with a time resolution of around 40-50 ms equivalent to a volume rate of 20-25 volumes per second. Measurements of RT3DE volumes will be performed off-line (4D analysis, TomTec Gmbh, Ubterschlessheim, Germany).

   For the study of MR, the standard color Doppler examination will be performed in the apical 4- and 2-chamber views to visualize the regurgitant jet; the flow convergence area will be recorded in the apical 4-chamber view in zoom mode, with color bar baseline set between 30 and 40 cm/s; finally, the CW Doppler tracing of the regurgitant jet will be acquired in the 4-chamber view.

   The PW Doppler examination will be performed positioning the sample volume at the level of the valve tips in the apical 4-chamber view for assessment of mitral inflow and at the level of the aortic anulus for assessment of aortic outflow.

   All conventional and TDI images will be acquired in a cineloop format during hold end-expiration (unless differently specified). Each cineloop and Doppler tracing will contain 3 cardiac cycles. All images and tracings will be stored on a CD-ROM for subsequent analysis. At the time of the echo examination blood pressure will be also measured.

   - Measurements. LV size will be evaluated measuring the end-diastolic and end-systolic diameters (EDD, ESD, cm) on 2D parasternal short-axis view images and calculating the end-diastolic and end-systolic volumes (EDV, ESV, ml) using RT3DE. The EDD and EDV will be indexed for body surface area. LV systolic function will be evaluated using both the ejection fraction (EF, %) calculated from volumes and the Doppler dP/dt (mmHg/ms) calculated from the CW MR tracing, when available. MR severity will be evaluated by: (1) the maximal regurgitant jet area visualized by color Doppler in the apical 4- and 2-chamber views (the average value of the two views will be calculated); (2) the PISA method; (3) the duration of the CW Doppler tracing of the regurgitant flow. Systolic pulmonary artery pressure (sPAP) will be calculated from the CW tricuspid regurgitation tracing.

   Several indexes of LV DYS have been selected based on published validation studies in which LV reverse remodeling has been considered as an end-point (single or combined) and at least 3 months of follow-up after CRT have been used. Dyssynchrony indexes will be calculated as previously reported in the literature (the respective cut-off value to predict positive response to CRT is shown in parentheses).

   M-mode indexes
   * Septal-to-posterior wall motion delay (cut-off value= 130 ms): measurement will be obtained from the M-mode tracing of the LV as the time interval between the maximal inward motion of the septum and the left posterior wall.
   * Lateral wall postsystolic displacement: difference of intervals from QRS onset to maximal systolic displacement of the basal LV lateral wall (assessed by M-mode in apical 4-chamber view) and from QRS onset to the beginning of the E wave (assessed by PW Doppler of mitral inflow); a positive value identifies a pathologic post-systolic contraction.

   TDI time intervals and indexes

   - Time to peak systolic velocity: the interval from onset of the QRS to the maximum positive velocity during the ejection period. The velocities in the isovolumic contraction and relaxation periods will not be used in this measurement. The region of interest (ROI) (6 x 6-mm circular shape) will be positioned in the middle of each segment. Time to peak velocity (Tv) will be measured on each curve from the beginning of the Q (or R)-wave on the ECG to the peak positive systolic velocity during the ejection phase, previously defined by the aortic valve opening and closure times. If a positive velocity will not be observed, the segment will be excluded from the calculation. If there will be multiple peaks in ejection period with the same velocity, the earliest peak will be chosen.
   * Time to peak velocity, including the postejection period: the interval from onset of the QRS to the maximum positive velocity, including the period after aortic valve closure. Everything else as above.
   * Time to peak strain: the interval from onset of the QRS to peak negative strain throughout the cardiac cycle, including postsystolic shortening. The region of interest (ROI) (6 x 12-mm oval shape) will be positioned in the middle of each segment. If negative strain will not be identified, the segment will be excluded from the calculation.
   * Time to peak strain exceeding aortic valve closure (ExcT: exceeding time): the interval between the marker of aortic closure and the nadir of the strain tracing. ExcT will be considered 0 when the nadir of strain curve will not exceed aortic valve closure. Everything else as above.

   In addition to the time intervals described above, the triplane TSI display of LV electro-mechanical delays will be evaluated visually (VT-TSI) during the systolic ejection phase to identify a severe lateral wall delay, marked by the presence of red color on the lateral wall (alone or in association with other severely delayed segments).

   Using the above described time intervals, the following DY indexes reported in the literature will be measured:
   * Septal-lateral delay (cut-off value= 65 ms): maximum time delay between peak systolic velocities among four basal segments in 4 chamber and 2 chamber view.
   * Anteroseptal-posterior delay (cut-off value= 65 ms): absolute time difference in time to peak systolic velocity, including the postejection period, between the basal inferolateral and basal anteroseptal segments.
   * Standard deviation in time to peak systolic velocity in the 12 basal and mid segments using both the two-dimensional tissue Doppler (cut-off value= 33.6 ms) and the novel triplane TSI modality (Tv-SD index).
   * Standard deviation in time to peak strain (cut-off value= 60 ms) among 12 basal and mid segments as a strain-derived dyssynchrony index (11).
   * Overall time of strain exceeding aortic valve closure (cut-off value= 760 ms) as the sum of 12 basal and mid segments ExcTs (10).

   Also, the combined approach based on the Tv-SD index (cut-off value= 34.4 ms) and VT-TSI severe lateral wall delay will be tested as described by Yu et al.

   RT3DE For each of the 16 LV segment, the time taken to reach the minimum regional volume will be measured and expressed as a percentage of the cardiac cycle. Then, the systolic dyssynchrony index (cut-off value= 8.3%) will be calculated as the standard deviation in time to minimum regional volume.

   Speckle-tracking analysis For each of the 6 segments of the mid-ventricle short-axis view, the time to peak radial strain will be measured. Then, the radial strain DYS (cut-off value= 130 ms) index will be calculated as the difference between earliest and latest time to peak strain.

   Echo core and peripheral laboratory. All investigators must obtain the approval of the core laboratory before participating in the study by sending a test CD-ROM of adequate quality to the core laboratory. The core laboratory will be located in Udine (L.P. Badano). A number of ultrasound images and tracings will be read in 2 peripheral laboratories to test the interlaboratory reproducibility for evaluation of dyssynchrony indexes.

   Optimization of atrio-ventricular delay will be performed at pre-discharge using Doppler echocardiography of transmitral flow to provide the maximum LV filling time without compromising cardiac resynchronization.

   Statistical analysis plan.
   * Descriptive statistics. Continuous variables will be described as mean and standard deviation and categorical variables as counts and percentages.
   * Statistical analysis: generality. The analysis for the continuous variables will be conducted by standard methods, unless there is evidence of important deviation from assumptions of normality, in which case non-parametric "bootstrap" methods will be used to generate confidence intervals. A two-sided p-value<0.05 will be considered statistically significant.

     1) Evaluation of feasibility and reproducibility of DYS indexes
   * Feasibility. Feasibility is defined for each DYS index by the number of patients in whom the index was actually measured or calculated relative to the number of patients in whom the measure or calculation was attempted. Feasibility will be evaluated separately in normals and in patients.
   * Measurements of DYS indexes will be repeated in 15 baseline normal studies and 15 baseline patient studies by the same and a second observer at least one week after the first assessment in the core laboratory to test intra and interobserver variability. The same normal and patient studies will be read in two peripheral laboratories to test the interlaboratory variability. All observers will be unaware of the patients' characteristics, including ECG data. The Lin correlation coefficient and the Bland-Altman limits of agreement (LOA) will be used to evaluate intraobserver, interobserver and interlaboratory variabilities.
   * To evaluate the strength of the association between dyssynchrony indexes values at baseline both in normals and in patients, the Pearson R and its 95% confidence interval (95% C.I.) will be computed.

     2) Evaluation of the effects of CRT
   * Variations over time. A paired Student t test or an exact symmetry homogeneity test will be used to compare baseline and 3-month continuous and categorical values, respectively.

     3) Evaluation of the predictive value of the dyssynchrony indexes
   * Association with CRT response and power analysis. The association between baseline dyssynchrony indexes, considered as continuous variables, and CRT response after 3 months will be assessed by means of a logistic model. With the available sample size and an alpha of 5%, the power for detecting the observed association of the dyssynchrony indexes with CRT response is computed to 80% for each parameter.
   * Association with CRT response based on DYS cut-off values. DYS parameters will also be dichotomized according to the pre-specified cut-off values derived from previous reports (see above). Model performances will be empirically compared through the c statistics for the discriminating ability (corresponding to the model based area under the ROC curve: the closer to 1, the better the model). Sensitivity and specificity of the dichotomized dyssynchrony parameters with respect to response will be computed.
   * Association with echocardiographic changes. The association of baseline dyssynchrony indexes on a continuous scale with the relative changes in echocardiographic EF and ESV after 3 months of CRT will be assessed by means of Pearson R.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Sinus rhythm.
* Chronic heart failure (>6 weeks duration) refractory to maximized drug therapy.
* NYHA class III-IV.
* LV ejection fraction less than 35% by RT3DE.
* Indexed LV end-diastolic diameter >3.2 cm/m2 by 2D echocardiography and/or indexed end-diastolic volume >75 ml/m2 by 3D echocardiography.

Exclusion Criteria:

* Hypertrophic, restrictive, obstructive cardiomyopathy.
* Primitive and hemodynamically significant valve disease (defined as valvular stenosis greater than mild, and 3+ or 4+/4+ valvular regurgitations).
* Constrictive pericarditis.
* Primitive pulmonary hypertension.
* Uncorrected congential heart disease.
* Patients candidate to heart surgery.
* Patients with acute myocardial infarction, severe unstable angina and stroke that occurred within 6 weeks prior the study enrollment.
* Patients with life expectation <1 year due to disease unrelated to the heart failure.
* Pregnant women.
* Refusal to give the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive consenting patients candidate to cardiac resynchronization therapy by clinical and electrocardiographic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2008-03; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Prediction of the combined end-point defined as NYHA class improvement by at least one grade and echocardiographic left ventricular end-systolic volume decrease by at least 10% with respect to baseline (variations are considered as relative values); | 3 months after biventricular pace-maker implant

SECONDARY OUTCOMES:
Feasibility and repeatibility of echocardiographic indexes of intraventricular dyssynchrony | 6 months
definition of reference values of echocardiographic mechanical dyssynchrony indexes in a population of healthy subjects; | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi P. Badano, M.D., Principal Investigator — Ospedale Universitario di Udine
Locations (1):
- Department of Cardiopulmonary Sciences - Ospedale Universitario, Udine, Italy

REFERENCES:
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Hawkins NM, Petrie MC, MacDonald MR, Hogg KJ, McMurray JJ. Selecting patients for cardiac resynchronization therapy: electrical or mechanical dyssynchrony? Eur Heart J. 2006 Jun;27(11):1270-81. doi: 10.1093/eurheartj/ehi826. Epub 2006 Mar 9. PMID 16527827
- [Background] Mollema SA, Bleeker GB, van der Wall EE, Schalij MJ, Bax JJ. Usefulness of QRS duration to predict response to cardiac resynchronization therapy in patients with end-stage heart failure. Am J Cardiol. 2007 Dec 1;100(11):1665-70. doi: 10.1016/j.amjcard.2007.06.071. Epub 2007 Oct 24. PMID 18036366
- [Background] Bax JJ, Abraham T, Barold SS, Breithardt OA, Fung JW, Garrigue S, Gorcsan J 3rd, Hayes DL, Kass DA, Knuuti J, Leclercq C, Linde C, Mark DB, Monaghan MJ, Nihoyannopoulos P, Schalij MJ, Stellbrink C, Yu CM. Cardiac resynchronization therapy: Part 1--issues before device implantation. J Am Coll Cardiol. 2005 Dec 20;46(12):2153-67. doi: 10.1016/j.jacc.2005.09.019. PMID 16360042
- [Background] Badano LP, Baldassi M, Ghio S, Mele D, Rigo F, Trambaiolo P, Fioretti PM. [Selection of patients undergoing cardiac resynchronization therapy: role of echocardiography]. G Ital Cardiol (Rome). 2006 Nov;7(11):724-38. Italian. PMID 17216914
- [Background] Yu CM, Abraham WT, Bax J, Chung E, Fedewa M, Ghio S, Leclercq C, Leon AR, Merlino J, Nihoyannopoulos P, Notabartolo D, Sun JP, Tavazzi L; PROSPECT Investigators. Predictors of response to cardiac resynchronization therapy (PROSPECT)--study design. Am Heart J. 2005 Apr;149(4):600-5. doi: 10.1016/j.ahj.2004.12.013. PMID 15990740
- [Background] Cleland JG, Abdellah AT, Khaleva O, Coletta AP, Clark AL. Clinical trials update from the European Society of Cardiology Congress 2007: 3CPO, ALOFT, PROSPECT and statins for heart failure. Eur J Heart Fail. 2007 Oct;9(10):1070-3. doi: 10.1016/j.ejheart.2007.09.005. Epub 2007 Sep 24. PMID 17890152
- [Background] Dohi K, Suffoletto MS, Schwartzman D, Ganz L, Pinsky MR, Gorcsan J 3rd. Utility of echocardiographic radial strain imaging to quantify left ventricular dyssynchrony and predict acute response to cardiac resynchronization therapy. Am J Cardiol. 2005 Jul 1;96(1):112-6. doi: 10.1016/j.amjcard.2005.03.032. PMID 15979447
- [Background] Suffoletto MS, Dohi K, Cannesson M, Saba S, Gorcsan J 3rd. Novel speckle-tracking radial strain from routine black-and-white echocardiographic images to quantify dyssynchrony and predict response to cardiac resynchronization therapy. Circulation. 2006 Feb 21;113(7):960-8. doi: 10.1161/CIRCULATIONAHA.105.571455. Epub 2006 Feb 13. PMID 16476850
- [Background] Porciani MC, Lilli A, Macioce R, Cappelli F, Demarchi G, Pappone A, Ricciardi G, Padeletti L. Utility of a new left ventricular asynchrony index as a predictor of reverse remodelling after cardiac resynchronization therapy. Eur Heart J. 2006 Aug;27(15):1818-23. doi: 10.1093/eurheartj/ehl133. Epub 2006 Jul 3. PMID 16818457
- [Background] Mele D, Pasanisi G, Capasso F, De Simone A, Morales MA, Poggio D, Capucci A, Tabacchi G, Sallusti L, Ferrari R. Left intraventricular myocardial deformation dyssynchrony identifies responders to cardiac resynchronization therapy in patients with heart failure. Eur Heart J. 2006 May;27(9):1070-8. doi: 10.1093/eurheartj/ehi814. Epub 2006 Mar 30. PMID 16574689
- [Background] Kapetanakis S, Kearney MT, Siva A, Gall N, Cooklin M, Monaghan MJ. Real-time three-dimensional echocardiography: a novel technique to quantify global left ventricular mechanical dyssynchrony. Circulation. 2005 Aug 16;112(7):992-1000. doi: 10.1161/CIRCULATIONAHA.104.474445. Epub 2005 Aug 8. PMID 16087800
- [Background] Marsan NA, Bleeker GB, Ypenburg C, Ghio S, van de Veire NR, Holman ER, van der Wall EE, Tavazzi L, Schalij MJ, Bax JJ. Real-time three-dimensional echocardiography permits quantification of left ventricular mechanical dyssynchrony and predicts acute response to cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2008 Apr;19(4):392-9. doi: 10.1111/j.1540-8167.2007.01056.x. Epub 2007 Dec 20. PMID 18179529
- [Background] Pitzalis MV, Iacoviello M, Romito R, Massari F, Rizzon B, Luzzi G, Guida P, Andriani A, Mastropasqua F, Rizzon P. Cardiac resynchronization therapy tailored by echocardiographic evaluation of ventricular asynchrony. J Am Coll Cardiol. 2002 Nov 6;40(9):1615-22. doi: 10.1016/s0735-1097(02)02337-9. PMID 12427414
- [Background] Sassone B, Capecchi A, Boggian G, Gabrieli L, Sacca S, Vandelli R, Petracci E, Mele D. Value of baseline left lateral wall postsystolic displacement assessed by M-mode to predict reverse remodeling by cardiac resynchronization therapy. Am J Cardiol. 2007 Aug 1;100(3):470-5. doi: 10.1016/j.amjcard.2007.02.107. Epub 2007 Jun 15. PMID 17659931
- [Background] Bax JJ, Bleeker GB, Marwick TH, Molhoek SG, Boersma E, Steendijk P, van der Wall EE, Schalij MJ. Left ventricular dyssynchrony predicts response and prognosis after cardiac resynchronization therapy. J Am Coll Cardiol. 2004 Nov 2;44(9):1834-40. doi: 10.1016/j.jacc.2004.08.016. PMID 15519016
- [Background] Gorcsan J 3rd, Kanzaki H, Bazaz R, Dohi K, Schwartzman D. Usefulness of echocardiographic tissue synchronization imaging to predict acute response to cardiac resynchronization therapy. Am J Cardiol. 2004 May 1;93(9):1178-81. doi: 10.1016/j.amjcard.2004.01.054. PMID 15110219
- [Background] Yu CM, Chau E, Sanderson JE, Fan K, Tang MO, Fung WH, Lin H, Kong SL, Lam YM, Hill MR, Lau CP. Tissue Doppler echocardiographic evidence of reverse remodeling and improved synchronicity by simultaneously delaying regional contraction after biventricular pacing therapy in heart failure. Circulation. 2002 Jan 29;105(4):438-45. doi: 10.1161/hc0402.102623. PMID 11815425
- [Background] Yu CM, Zhang Q, Fung JW, Chan HC, Chan YS, Yip GW, Kong SL, Lin H, Zhang Y, Sanderson JE. A novel tool to assess systolic asynchrony and identify responders of cardiac resynchronization therapy by tissue synchronization imaging. J Am Coll Cardiol. 2005 Mar 1;45(5):677-84. doi: 10.1016/j.jacc.2004.12.003. PMID 15734610
- [Background] Butter C, Wellnhofer E, Seifert M, Schlegl M, Hoersch W, Goehring A, Fleck E. Time course of left ventricular volumes in severe congestive heart failure patients treated by optimized AV sequential left ventricular pacing alone--a 3-dimensional echocardiographic study. Am Heart J. 2006 Jan;151(1):115-23. doi: 10.1016/j.ahj.2005.02.047. PMID 16368302